CLINICAL TRIAL: NCT04861818
Title: The Role of the Time of Day in the Effects of Exercise on Memory in Heathy Young Adults
Acronym: TEEMY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20-0141
Record Dates: First submitted 2020-03-23; First posted 2021-04-27 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Aerobic Exercise; Cognitive Change
Keywords: Aerobic exercise; Physical activity; Cognition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning group (Experimental): Participant are assigned to the morning group (7-9am) for 30-min exercise/rest interventions.
  Interventions: Behavioral: Moderate-intensity aerobic exercise
- Afternoon group (Experimental): Participant are assigned to the afternoon group (3-5pm) for 30-min exercise/rest interventions.
  Interventions: Behavioral: Moderate-intensity aerobic exercise

INTERVENTIONS:
Behavioral: Moderate-intensity aerobic exercise — Eligible participants will come into the lab on day 1 and 3 at the same time of day (either morning at 7-10am or afternoon at 3-5pm). They will be then randomly assigned for a rest or an exercise session prior to the memory test. For the rest condition, they will be required to sit and relax while watching Planet Earth for 30 minutes on a cycle ergometer. During the exercise session, they will complete a moderate-intensity cardiovascular exercise for 20 minutes following a 5-min warm-up and followed by a 5-min cool-down on a cycle ergometer. They will start the memory test immediately after the rest/exercise session.

SUMMARY:
Cumulative evidence indicates that a single bout of exercise has beneficial impacts on memory in young adults. From a physiological perspective, acute exercise leads to changes of heart rate variability (HRV), which is associated with memory retrieval process. From a psychological perspective, acute exercise increases the arousal level and thus facilitates cognitive processing including memory storage and retrieval. Such HRV- and/or arousal-based effects of exercise on memory could be differed by the time of day in young adults based on their circadian rhythms of HRV. Moreover, young adults prefer afternoon or evening to morning in their circadian rhythms, demonstrating less wakefulness and lower memory performance in the morning relative to afternoon. Based on the potential psychophysiological mechanisms, exercise could impact young adults' memory differently by the time of day. The investigators aim to 1) determine the extent to which the time of day modulates how moderate-intensity cardiovascular exercise impacts verbal-auditory and visuospatial short- and long-term memory in young adults, and 2) consider potential psychological and physiological markers that may mediate exercise's effects on cognitive performance. As cognitive benefits of exercise might differ by the time of day, it is important to investigate such interaction and make the right recommendations of the timing of exercise for young adults in academic settings.

DETAILED DESCRIPTION:
Cumulative evidence indicates that a single bout of exercise has beneficial impacts on short- and long-term memory in young adults. From a physiological perspective, acute exercise leads to changes of heart rate variability (HRV), which is associated with memory retrieval process. From a psychological perspective, acute exercise increases the arousal level and thus facilitates cognitive processing including memory storage and retrieval. Such HRV- and/or arousal-based effects of exercise on memory could be differed by the time of day in young adults based on their circadian rhythms of HRV; sleep-wake transition led to rapid changes of HRV. Moreover, young adults prefer afternoon or evening to morning, showing less wakefulness and lower memory performance in the morning relative to afternoon. Based on the potential physiological and/or psychological mechanisms, exercise could impact young adults' memory differently by the time of day. Few studies, however, tested the effects of exercise on memory based on the time of day; rather, a recent study found null effects of exercise-induced arousal on implicit and explicit memory performance in college students in the morning.

The investigators here aim to 1) determine the extent to which the time of day moderates how moderate-intensity cardiovascular exercise impacts verbal-auditory and visuo-spatial short- and long-term memory in young adults, and 2) consider potential physiological and psychological markers that may mediate exercise's effects on cognitive performance. Specifically, the investigators will conduct a mixed-design randomized experiment to compare the effects of a single session of moderate-intensity cardiovascular exercise on cognitive performance at two times of day - in the morning (7 - 9 AM) and late afternoon (3 - 5 PM). Participants in each of two groups (morning versus afternoon) will complete two sessions of cognitive tests - at baseline without exercise and after an exercise intervention, while their emotional states, arousal levels, and heart rate (HR) will be measured at baseline, before, during, and after the exercise and memory sessions. The hypotheses are 1) acute exercise in the morning will be more beneficial for short- and long-term memory than an equal volume of exercise in the afternoon; 2) resting HRV and changes in perceived arousal and emotional states will be associated with memory performance following the exercise intervention. The rationale for the hypotheses is that cognitive benefits of exercise can differ by the preference for the time of day, so it is important to investigate such interactions to inform recommendations of the timing of exercise for young adults in academic settings. Moreover, exploring the role of psychophysiological markers in mediating exercise effects on cognition help to further understanding of the benefits of exercise for brain health.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-25.
* Currently meeting the American College of Sports Medicine's recommended guidelines of activity (at least 90 min/week of moderate and/or vigorous physical activity).
* Willing to participate for 4 days (2 visits) and refrain from exercise outside of the lab for 4 days (1 day before and the day of two visits).

Exclusion Criteria:

* Any known history of cardiac, pulmonary, or metabolic disease (e.g. cardiovascular disease, asthma, diabetes).
* A current musculoskeletal injury, mental illness (e.g., depression, anxiety, or stress disorders), or sleep disorder.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Verbal episodic memory change | Immediately after the intervention, the first cognitive test
  Verbal episodic memory will be assessed immediately and 24 hour after intervention (rest and exercise) using the Auditory Verbal Learning Test (AVLT trial 1 - 8; max/min score: 15/0 for each trial)
Visual episodic memory change | Immediately after the intervention, the second cognitive test
  Verbal episodic memory will be assessed immediately after intervention (rest and exercise) using the NIH Toolbox Picture Sequence Memory Test (max/min score: 30/0).
Lure discrimination index change | Immediately after the intervention, the third cognitive test
  Lure discrimination index will be assessed immediately after intervention (rest and exercise) using the Mnemonic Similarity Task (max/min score: 1/0).
Working memory change | Immediately after the intervention, the fourth cognitive test
  Verbal episodic memory will be assessed immediately after intervention (rest and exercise) using the Digits Span Forward and Backward Task (max/min score: 14/0).

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Shin Park, PhD, Principal Investigator — UNC Greensboro
Locations (1):
- UNC Greensboro, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No